CLINICAL TRIAL: NCT05319886
Title: A Phase IV Observational Study Evaluating the Efficacy and Safety of Anlotinib in Combination With Penpulimab as First-line Treatment in Elderly Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Observational Study of the Efficacy and Safety of Anlotinib Combined With Penpulimab in Elderly Lung Cancer Patients
Acronym: AP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: LC202103001
Record Dates: First submitted 2022-04-01; First posted 2022-04-08 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Lung Cancer; Lung Carcinoma; Non Small Cell Lung Cancer; Non-small Cell Carcinoma; Lung Neoplasm
Keywords: Anlotinib; Penpulimab
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — anlotinib; penpulimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anlotinib and Penpulimab
  Interventions: Drug: Anlotinib and Penpulimab

INTERVENTIONS:
Drug: Anlotinib and Penpulimab — Anlotinib 12mg, po, qd, with 2 weeks off for 1 week. Penpulimab 200mg, ivgtt, q3w. Efficacy was evaluated every 2 cycles. Efficacy evaluation was performed every 2 cycles during the follow-up study. Patients with disease control (CR+PR+SD) and tolerable adverse reactions continued to take the drug until the investigator considered that the patient was not suitable to continue the drug or the efficacy was evaluated as PD. Safety evaluations were performed concurrently with the dosing period. No other antitumor therapy can be administered until PD.
  Other Names: AL3818 and AK105

SUMMARY:
This prospective observational study will evaluate the efficacy and safety of anlotinib in combination with Penpulimab in elderly patients with lung cancer. Data will be collected from each patient at baseline and after 4-6 cycles of therapy.

DETAILED DESCRIPTION:
This research study is a Phase IV clinical trial. Participants are being involved in the portion of the study to observe the efficacy and safety of an observational intervention and also tries to evaluate the disease control rate (such as Progression-Free-Survival, overall survival, Objective Response Rate, Disease control rates, Duration of Response, Quality of Life and Adverse events).

Anlotinib is a small molecule multi-target tyrosine kinase inhibitor, can effectively inhibit VEGFR, PDGFR, FGFR, c-Kit and other kinases, with anti-tumor angiogenesis and tumor growth inhibiting effects. Penpulimab injection is a new PD-1 monoclonal antibody drug, was approved for marketing by the State Drug Administration (NMPA) of China for the indication: treatment of adult patients with relapsed or refractory classic Hodgkin's lymphoma (r/r cHL) who have undergone at least second-line systemic chemotherapy. By putting these two drugs together, the investigators hope that it will have a greater effect on cancer growth in elderly patients with lung cancer.

Efficacy evaluation was performed every 2 cycles during the follow-up study. Patients with disease control (complete response (CR)+partial response (PR)+stable disease (SD)) and tolerable adverse reactions continued to take the drug until the investigator considered that the patient was not suitable to continue the drug or the efficacy was evaluated as disease progression (PD). Safety evaluations were performed concurrently with the dosing period. No other antitumor therapy can be administered until PD.

The purpose of this study is to:

* Test the efficacy of these two drugs Anlotinib and Penpulimab in elderly lung cancer;
* Determine the Progression-Free-Survival of the combination;
* Further evaluate the side effect profile for the combination of Anlotinib and Penpulimab in elderly lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* At least 65 years old;
* Non-small cell lung cancer with locally advanced, recurrent or metastasis, which confirmed by histologically or cytologically (except sputum cytology) and evaluated as IIIB-IV stage, who are unresectable or unable to undergo radical radiotherapy or refuse radical radiotherapy. (If multiple tumor components are mixed, it should be classified according to their predominant cell type);
* Participants are required to have one measurable disease per RECIST 1.1;
* Unsuitable or unwilling to receive radical treatment methods (such as radical chemoradiotherapy and/or surgery) and have not received prior systemic therapy;
* ECOG performance status of 0 to 2; The expected survival is more than 3 months;
* Adequate organ and marrow function defined as follows:

  * Hemoglobin (HB) ≥90 g/L (no blood transfusion within 28 days);
  * Absolute neutrophil count (ANC) ≥1.5×109/L;
  * Platelet count (PLT) ≥ 100×109/L;
  * Aspartate Transaminase (AST) ≤ 1.5 x upper limit of normal (ULN);
  * Alaninetransaminase (ALT) ≤ 1.5 x ULN (ALT and AST ≤ 5 x ULN if liver metastases are present);
  * Alkaline phosphatase (ALP) ≤ 1.5 x ULN;
  * Albumin (ALB) ≥ 30g/L;
  * Creatinine ≤1.5 x ULN or Creatinine Clearance (CCr) ≥ 60 ml/min;
  * International normalized ratio (INR) ≤ 1.5 x ULN;
  * Partial thromboplastin time (APTT) ≤ 1.5 x ULN;
  * Prothrombin time (PT) ≤ 1.5 x ULN ;
  * Thyrotropic hormone (TSH) ≤ ULN (When TSH value is abnormal, T3 and T4 levels is normal, which can be enrolled);
  * Urine protein < (++), or 24-hour urine protein amount < 1.0 g ;
  * Patients must have adequate cardiac function, defined as:

Left ventricular ejection fraction (LVEF) > 50% as determined by cardiac echocardiogram.

-Patients enrolled in this study voluntarily and signed an informed consent with a good compliance.

Exclusion Criteria:

* Participants who have active infection;
* Patients with known immunodeficiency diseases (e.g. psoriasis, active arthritis, immune nephropathy, HIV, etc);
* Participants with no measurable disease;
* Patients with cancerous meningitis and spinal cord compression;
* Participants with active central nervous system (CNS) metastases (clinically stable and maintained for at least 2 weeks after adequate treatment of CNS metastases and do not require treatment such as glucocorticoids and dehydrating drugs are eligible for enrollment);
* Previously treated with chemotherapy drugs (except neoadjuvant therapy) / targeted drugs / immunotherapy;
* Participants who were confirmed severe abnormalities of gastrointestinal function (e.g. inability to take oral medications, uncontrollable nausea or vomiting, history of major gastrointestinal resection, untreated recurrent diarrhea, untreated gastric disease requiring long-term acid-suppressing PPI-like medications, Crohn's disease, ulcerative colitis);
* Patients with central squamous lung cancer on imaging;
* Patients who had an arterial/venous thrombotic event within 6 months, such as cerebrovascular accident (temporary ischemic attack is excluded), deep vein thrombosis and pulmonary embolism;
* Patients whose imaging shows that the tumor has invaded a significant vessel or have a high risk of fatal hemorrhage due to tumor invasion of a significant vessel during the follow-up study judged by the investigator; or who have bleeding tendencies (e.g., active peptic ulcer) or receiving thrombolytic or anticoagulant therapy such as warfarin, heparin, or their analogs;
* Patients who had antineoplastic therapy against other malignancies, including radiotherapy, chemotherapy, immunotherapy and herbal medicine (except previously eradicated malignancies without recurrent metastases for ≥ 5 years);
* Patients with uncontrollable pleural effusion, pericardial effusion or ascites requiring repeated drainage (except patients who do not require drainage of effusion or whose effusion does not increase significantly after 3 days of cessation of drainage);
* Patients who have used immunosuppressive drugs within 4 weeks prior to the study treatment, except for topical glucocorticoids by nasal spray, inhalation or other routes or physiologic doses of systemic glucocorticoids (no more than 10 mg/day of prednisone or equivalent doses of other glucocorticoids);
* Patients who have known or suspected active autoimmune disease (congenital or acquired), such as interstitial pneumonia, uveitis, enterocolitis, hepatitis, pituitary inflammation, vasculitis, nephritis, thyroiditis, etc. (Patients with vitiligo or asthma that has completely resolved in childhood and does not require any intervention in adulthood may be enrolled; Patients with type I diabetes with good insulin control may be enrolled);
* Patients who have known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
* Anticipants who have hypersensitivity to any component of anlotinib and monoclonal antibodies;
* Anticipants who have active interstitial lung disease requiring treatment;
* Anticipants who have a history of psychotropic substance abuse and are unable to abstain or have a psychiatric disorder;
* Anticipants who have participated in another anti-tumor clinical trial within four weeks;
* Anticipants who administered anti-infective vaccines (e.g., influenza virus vaccine, human papillomavirus vaccine) within 4 weeks prior to study therapy; During the treatment period, in addition to inactive vaccines, other vaccines are prohibited;
* Anticipants who have undergone major surgery (except for diagnostic purposes) within 4 weeks (28 days) prior to the administration of the study;
* Patients who are not suitable for enrollment in the judgment of the investigator.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: At least 65 years old with locally advanced, recurrent or metastatic stage IIIB-IV non-small cell lung cancer.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 2 years
  The time from the start of treatment until objective tumor progression or death. For participants who don't show progression or die until the end of treatment, the date of last contact is taken as the censoring time.

SECONDARY OUTCOMES:
Overall Survival | 2 years
  Overall survival is the time elapsed between enrollment and death of any cause. For participants who don't die until the end of treatment, the overall survival data will be analyzed retrospectively based on their date of death after the end of study.
Objective Response Rate | 2 years
  This refers to the percentage of patients with a certain amount of tumor shrinkage that is maintained for a certain period of time, including CR and PR.
Disease control rates | 2 years
  Includes the number of cases of CR, PR, and SD with confirmed disease as a percentage of patients evaluable for efficacy.
Duration of Response | 2 years
  Time between the start of the first evaluation of the tumor as CR or PR and the first evaluation of PD or death from any cause
Adverse events | 2 years
  An adverse event is any untoward medical occurrence in a patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided